CLINICAL TRIAL: NCT03120975
Title: Improvement of Antibiotic Use in Hospitals Through Pragmatic, Multifaceted, Computerized Interventions: a Multicentre, Cluster-randomized Trial - COMPASS Study (COMPuterized Antibiotic Stewardship Study)
Brief Title: Computerized Antibiotic Stewardship Study
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benedikt Huttner (Other)
Collaborators: Swiss National Science Foundation (Other); University of Geneva, Switzerland (Other); Ente Ospedaliero Cantonale, Ticino, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Benedikt Huttner, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-00454; 407240_167079 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Communicable Diseases
Keywords: Anti-Infective Agents; Decision Support Systems, Clinical; Quality Improvement
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Parallel group, cluster-randomized superiority trial
Who Masked: Outcomes Assessor
Masking Description: Masking for care providers and investigators is unfortunately not feasible. Outcome assessors and data analysts will be blinded to the study arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized decision support (Experimental)
  Interventions: Other: Computerized decision support and audit & feedback; Other: Audit & Feedback; Other: Standard antibiotic stewardship
- Standard antibiotic stewardship (Active Comparator)
  Interventions: Other: Standard antibiotic stewardship

INTERVENTIONS:
Other: Computerized decision support and audit & feedback — * suggestion of guideline concordant antimicrobial treatment based on indication entry in the computerized physician order entry system
  * mandatory reevaluation of antimicrobial therapy therapy on calendar day 4 of treatment
  * suggestion of standard antimicrobial treatment duration according to indication
  Arms: Computerized decision support
Other: Audit & Feedback — * regular (at least monthly) feedback of antibiotic use quality indicators (on the ward level)
  Arms: Computerized decision support
Other: Standard antibiotic stewardship — * Infectious diseases consultation "on demand"
  * Review of positive blood cultures
  * Availability of a antibiotic use guidelines (on paper and as PDF)

SUMMARY:
Prescribing antibiotics frequently poses problems in practice, since patients don't always receive the right dosage of the right antibiotic for the right period of time. This promotes the emergence and spread of antibiotic resistance. The investigators of this trial aim to develop a system designed to help doctors to use antibiotics more appropriately. Under COMPASS (COMPuterized Antibiotic Stewardship Study), doctors in three Swiss hospitals will receive tips on the use of antibiotics that are integrated directly into electronic health record and will also be given regular feedback on their use of antibiotics. Parallel to this, data on the antimicrobial prescription practices of a control group which is not using the system will be collected.

DETAILED DESCRIPTION:
Inappropriate use of antimicrobials favours the spread and emergence of antimicrobial resistance and other adverse patient outcomes. Antimicrobial stewardship (AMS) programs aim to promote the appropriate use of antimicrobials. Most AMS interventions are based on manual, personalized peer review of antibiotic prescriptions by specialists and are therefore time and resource intensive. Informatics based, computerized approaches to AMS are a promising way to "automatize" AMS, but there have been only few randomized controlled trials analysing their effectiveness in the hospital setting.

The primary research question of this study is whether a multi-modal, computerized antibiotic stewardship intervention (I) reduces overall antibiotic exposure (O) in adult patients hospitalized in acute-care wards of secondary and tertiary care centers (P) compared to no such intervention ("standard-of- care") (C) over a one year time period (T) (the letters refer to the corresponding constituents of the PICOT framework).

The primary objective of the study is to use the methodological rigor of a parallel group, cluster-randomized, controlled superiority trial in three Swiss hospitals to answer the primary research question. Secondary objectives are to assess the impact of the intervention on quality of antibiotic use, patient, microbiologic and economic outcomes.

The primary outcome will be the difference in overall systemic antibiotic use measured in days of therapy (DOT) per admission based on administration data recorded in the electronic health record (EHR) over the whole intervention period. Secondary outcomes will include qualitative and quantitative antimicrobial use indicators (including non-HIV antivirals and antifungals), economic outcomes and key clinical and microbiologic indicators and patient safety indicators such as changes in readmission rates, need for intensive care and mortality.

The study hypothesis is that the multimodal intervention is superior to standard-of-care regarding the primary outcome, i.e. that the intervention leads to a statistically significant reduction in overall antibiotic use expressed as days of therapy per admission compared to no such intervention ("standard-of-care" antibiotic stewardship).

ELIGIBILITY:
Inclusion Criteria:

CLUSTER (WARD) LEVEL

* Acute-care wards with at least 150 admissions/year
* Use of a computerized physician order entry system (CPOE)

PHYSICIAN LEVEL * All physicians involved in antibiotic prescribing decisions in the participating wards

PATIENT LEVEL

* All patients hospitalized in the participating wards

Exclusion Criteria:

CLUSTER (WARD) LEVEL

* Emergency room
* Outpatient clinics
* Overflow wards
* Absence of a matchable wards with regard to specialty and baseline antibiotic use
* Hematopoietic stem cell

PHYSICIAN LEVEL * None

PATIENT LEVEL

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16176 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Days of therapy (DOT)/admission | 12 months
  Overall days of therapy of antibiotics per admission on the ward level

SECONDARY OUTCOMES:
Days of therapy(DOT)/100 patient days | 12 months
  Overall days of therapy per 100 patient days (PD) on the ward level
Defined daily doses (DDD)/100 patient days (PD) and per admission | 12 months
  Overall defined daily doses per 100 patient days and admission on the ward level
Antimicrobial days (AD) per 100 PD and per admission | 12 months
  Length of therapy per 100 PD and per admission
Days per treatment period overall | 12 months
  Overall days per treatment period. A treatment period is defined as antibiotic treatment not interrupted by more than one calendar day or discharge.
30 day-mortality | 12 months
  All cause 30 day-mortality
In-hospital mortality | 12 months
  All-cause in-hospital mortality
Hospital readmission within 30 days of discharge | 12 months
  Unplanned hospital readmission within 30 days of discharge
Hospital length of stay (LOS) | 12 months
  Hospital length of stay
ICU transfer | 12 months
  % of admissions transferred to ICU after initial non-ICU admission
Guideline compliance | 12 months
  Proportion of patients treated in compliance with facility-based guideline
De-escalation | 12 months
  Proportion of patients with "de-escalation" and "escalation" of antibiotic therapy by calendar day 4 of treatment
IV-oral switch | 12 months
  Proportion of patients converted from intravenous to oral therapy between days 4 and 7
appropriate diagnostic exams | 12 months
  proportion of patients with appropriate diagnostic exams
Incidence of Clostridium difficile infections (CDI) | 12 months
  Incidence of healthcare-facility onset Clostridium difficile infection denominated by 10 000 PD and admission
Incidence of multidrug-resistant organisms (MDRO) | 12 months
  Incidence of clinical cultures with multidrug resistant organisms (methicillin-resistant Staphylococcus aureus (MRSA), Extended spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E), carbapenemase-producing Enterobacteriaceae (CPE), vancomycin-resistant enterococci (VRE), multidrug resistant P. aeruginosa) denominated per 1000 PD and admissions
User satisfaction | 12 months
  User satisfaction with the system
Costs of administered antimicrobials | 12 months
  Costs of administered antimicrobials (overall and by class) per admission and per admission receiving antibiotics
costs of the intervention | 12 months
  total costs of the intervention
number of infectious diseases consultations | 12 months
  proportion of patients with infectious diseases consultation
Days per treatment period for community acquired pneumonia | 12 months
  A treatment period is defined as antibiotic treatment not interrupted by more than one calendar day or discharge.
Days per treatment period for upper urinary tract infection | 12 months
  A treatment period is defined as antibiotic treatment not interrupted by more than one calendar day or discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt D Huttner, MD, MS, Principal Investigator — Geneva University Hospitals and University of Geneva
Locations (3):
- Switzerland (3):
  - Geneva University Hospitals, Geneva, Canton of Geneva
  - Ente Ospedaliera Cantonale - Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Ente Ospedaliera Cantonale - Ospedale Civico, Lugano, Canton Ticino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catho G, De Kraker M, Waldispuhl Suter B, Valotti R, Harbarth S, Kaiser L, Elzi L, Meyer R, Bernasconi E, Huttner BD. Study protocol for a multicentre, cluster randomised, superiority trial evaluating the impact of computerised decision support, audit and feedback on antibiotic use: the COMPuterized Antibiotic Stewardship Study (COMPASS). BMJ Open. 2018 Jun 27;8(6):e022666. doi: 10.1136/bmjopen-2018-022666. PMID 29950480
- [Result] Catho G, Centemero NS, Catho H, Ranzani A, Balmelli C, Landelle C, Zanichelli V, Huttner BD; on the behalf of the Q-COMPASS study group. Factors determining the adherence to antimicrobial guidelines and the adoption of computerised decision support systems by physicians: A qualitative study in three European hospitals. Int J Med Inform. 2020 Sep;141:104233. doi: 10.1016/j.ijmedinf.2020.104233. Epub 2020 Jul 13. PMID 32736330
- [Derived] Catho G, Sauser J, Coray V, Da Silva S, Elzi L, Harbarth S, Kaiser L, Marti C, Meyer R, Pagnamenta F, Portela J, Prendki V, Ranzani A, Centemero NS, Stirnemann J, Valotti R, Vernaz N, Suter BW, Bernasconi E, Huttner BD; COMPASS study group. Impact of interactive computerised decision support for hospital antibiotic use (COMPASS): an open-label, cluster-randomised trial in three Swiss hospitals. Lancet Infect Dis. 2022 Oct;22(10):1493-1502. doi: 10.1016/S1473-3099(22)00308-5. Epub 2022 Jul 20. PMID 35870478
- See also: Lay summary of the project — http://www.nfp72.ch/en/projects/module-3-optimised-use-of-antibiotics/using-computers-to-improve-prescription-practices